CLINICAL TRIAL: NCT03083665
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter, Parallel-group Study to Evaluate the Efficacy and Safety of Adjunctive Brivaracetam in Subjects (>=16 to 80 Years of Age) With Partial Seizures With or Without Secondary Generalization
Brief Title: A Study to Evaluate the Efficacy and Safety of Brivaracetam in Study Participants (>=16 to 80 Years of Age) With Epilepsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EP0083
Record Dates: First submitted 2017-02-28; First posted 2017-03-20 (Actual); Results first posted 2023-11-09 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Partial Seizures With or Without Secondary Generalization; Epilepsy
Keywords: Epilepsy; Partial seizures with or without secondary generalization; Brivaracetam; Briviact
MeSH Terms: conditions — Epilepsy | interventions — brivaracetam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): * 12 weeks Treatment Period: Subjects will receive Placebo
  * 4 weeks Down-Titration Period: Subjects will receive Placebo
  Interventions: Drug: Placebo
- BRV 50 mg/day (Experimental): 12 weeks Treatment Period: Subjects will receive BRV 50 mg/day
  - Subjects entering into the Long term follow up (LTFU) study or managed access program (MAP): 2 weeks Transition Period: Subjects will receive BRV 50 mg/day followed by LTFU or MAP: Subjects will receive BRV 100 mg/day
  - Subjects not entering into the LTFU study or MAP: 4 weeks Down-Titration Period: Subjects will receive BRV 25 mg/day for 1 week followed by Placebo for 3 weeks, followed by a Study Drug-Free Period
  Interventions: Drug: Placebo; Drug: Brivaracetam
- BRV 200 mg/day (Experimental): 12 weeks Treatment Period: Subjects will receive BRV 200 mg/day
  - Subjects entering into the Long term follow up (LTFU) study or managed access program (MAP): 2 weeks Transition Period: Subjects will receive BRV 150 mg/day followed by LTFU or MAP: Subjects will receive BRV 100 mg/day
  - Subjects not entering into the LTFU study or MAP: 4 weeks Down-Titration Period: Subjects will receive BRV 150 mg/day for 1 week followed by BRV 100 mg/day for 1 week, followed by BRV 50 mg/day for 1 week, followed by BRV 25 mg/day for 1 week followed by a Study Drug-Free Period
  Interventions: Drug: Placebo; Drug: Brivaracetam

INTERVENTIONS:
Drug: Placebo — * Pharmaceutical form: Film-coated tablets
  * Route of administration: Oral use
Drug: Brivaracetam — * Pharmaceutical form: Film-coated tablets
  * Concentration: 25 mg tablets and 50 mg tablets
  * Route of administration: Oral use
  Other Names: Briviact
  Arms: BRV 200 mg/day; BRV 50 mg/day

SUMMARY:
The purpose of the study is to evaluate the efficacy of brivaracetam (BRV) compared to placebo (PBO) as adjunctive treatment in subjects (>=16 to 80 years of age) with partial seizures with or without secondary generalization despite current treatment with 1 or 2 concomitant antiepileptic drugs (AEDs) and to assess the safety and tolerability of BRV in subjects >= 16 years to 80 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Subjects (male or female) from 16 to 80 years of age at Visit 1, both inclusive
* Female subjects with childbearing potential are eligible if they use a medically accepted contraceptive method
* Subjects having at least 8 partial seizures (according to the 1981 ILAE classification) during the 8-Week Baseline Period with at least 2 partial seizures during each 4-week interval of the Baseline Period
* Subjects having at least 2 partial seizures whether or not secondary generalization per month during the 3 months preceding Visit 1
* Subjects uncontrolled while treated by 1 or 2 permitted concomitant antiepileptic drug [AED](s). Vagal Nerve Stimulation (VNS) is allowed and will be counted as a concomitant AED

Exclusion Criteria:

* Subject has history or presence of status epilepticus during the year preceding Visit 1 or during Baseline
* Subject is currently treated with levetiracetam
* Subject has taken levetiracetam within 90 days prior to Visit 1

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 449 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (94):
- China (23):
  - Ep0083 905, Beijing
  - Ep0083 906, Beijing
  - Ep0083 907, Changchun
  - Ep0083 901, Chengdu
  - Ep0083 902, Guangzhou
  - Ep0083 909, Guangzhou
  - Ep0083 917, Guangzhou
  - Ep0083 920, Guangzhou
  - Ep0083 922, Guangzhou
  - Ep0083 924, Guangzhou
  - Ep0083 912, Hangzhou
  - Ep0083 908, Lanzhou
  - Ep0083 921, Nanchang
  - Ep0083 926, Pingxiang
  - Ep0083 910, Shijiazhuang
  - Ep0083 925, Suzhou
  - Ep0083 913, Wenzhou
  - Ep0083 927, Xi'an
  - Ep0083 930, Xinxiang
  - Ep0083 916, Yinchuan
  - Ep0083 918, Zhanjiang
  - Ep0083 904, Zhengzhou
  - Ep0083 923, Zunyi
- Japan (40):
  - Ep0083 148, Adachi-ku
  - Ep0083 116, Asaka
  - Ep0083 126, Bunkyō City
  - Ep0083 127, Bunkyō City
  - Ep0083 146, Chiba
  - Ep0083 122, Hachinohe
  - Ep0083 111, Hamamatsu
  - Ep0083 141, Higashisonogi-gun Kawatana-cho
  - Ep0083 110, Hiroshima
  - Ep0083 121, Itami
  - Ep0083 102, Kagoshima
  - Ep0083 142, Kamakura
  - Ep0083 140, Kawasaki
  - Ep0083 123, Kodaira
  - Ep0083 115, Kokubunji
  - Ep0083 132, Kōriyama
  - Ep0083 112, Kōshi
  - Ep0083 128, Kurume
  - Ep0083 124, Kyoto
  - Ep0083 147, Kyoto
  - Ep0083 105, Nagakute
  - Ep0083 118, Nagoya
  - Ep0083 136, Nagoya
  - Ep0083 117, Nara
  - Ep0083 129, Neyagawa
  - Ep0083 106, Niigata
  - Ep0083 130, Ôsaka
  - Ep0083 131, Ōtsu
  - Ep0083 114, Saitama
  - Ep0083 101, Sapporo
  - Ep0083 103, Sendai
  - Ep0083 144, Shinjuku-ku
  - Ep0083 104, Shizuoka
  - Ep0083 108, Suita
  - Ep0083 137, Suita
  - Ep0083 138, Tsukuba
  - Ep0083 133, Ushiku
  - Ep0083 109, Yamagata
  - Ep0083 120, Yokohama
  - Ep0083 150, Yokohama
- Malaysia (8):
  - Ep0083 207, Kota Bharu
  - Ep0083 201, Kuala Lumpur
  - Ep0083 206, Kuala Terengganu
  - Ep0083 204, Kuching
  - Ep0083 209, Miri
  - Ep0083 202, Perai
  - Ep0083 208, Pulau Pinang
  - Ep0083 203, Sungai Buloh
- Philippines (8):
  - Ep0083 303, Cebu City
  - Ep0083 304, Cebu City
  - Ep0083 306, Davao City
  - Ep0083 307, Iloilo City
  - Ep0083 301, Manila
  - Ep0083 302, Manila
  - Ep0083 310, Manila
  - Ep0083 309, Quezon City
- Singapore (2):
  - Ep0083 401, Singapore
  - Ep0083 402, Singapore
- Taiwan (5):
  - Ep0083 502, Chiayi City
  - Ep0083 505, Kaohsiung City
  - Ep0083 503, Taichung
  - Ep0083 504, Taichung
  - Ep0083 501, Tainan
- Thailand (8):
  - Ep0083 602, Bangkok
  - Ep0083 605, Bangkok
  - Ep0083 606, Bangkok
  - Ep0083 607, Bangkok
  - Ep0083 609, Bangkok
  - Ep0083 601, Khon Kaen
  - Ep0083 603, Muang
  - Ep0083 608, Muang

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: https://vivli.org/

REFERENCES:
- [Result] Usui N, Zhou D, Qin B, Tiamkao S, Cabral-Lim L, Lim KS, Lim SH, Tsai JJ, Watanabe J, Sun W, Dickson N, Moseley B, Bourikas D, Inoue Y. Temporal Profile of Treatment-Emergent Adverse Events in Adult Asian Patients with Focal-Onset Seizures During Adjunctive Brivaracetam Treatment: Post Hoc Analysis of a Phase 3, Randomized Trial. Adv Ther. 2025 Nov;42(11):5639-5652. doi: 10.1007/s12325-025-03357-7. Epub 2025 Sep 13. PMID 40944847

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in August 2017 and concluded in June 2022.
Pre-assignment Details: The Participant Flow refers to the Randomized Set. Double-Blind Period included Treatment Period and the Down-Titration Period plus Study Drug-Free Period or the Transition Period.
Groups:
- Placebo: Participants received matching Placebo as film-coated tablets, administered orally, twice daily (bid), during 12 weeks of Treatment Period. At the end of the Treatment Period, participants who entered long-term follow-up (LTFU) study (EP0085 (NCT03250377)) or managed access program (MAP), the same matching Placebo dose was kept during 2 weeks of Transition Period and brivaracetam (BRV) 100 milligrams/day (mg/day) in LTFU study or MAP. Participants who did not enter the LTFU study or MAP had 4 weeks Down-Titration Period followed by a Study Drug-Free Period (no drug for 2 weeks). During Down-Titration Period, participants received the same Placebo dose for 4 weeks.
- BRV 50 mg/Day: Participants received BRV 50 mg/day as film-coated tablets, administered orally, bid, during 12 weeks of Treatment Period. At the end of the Treatment Period, participants who entered the LTFU study or MAP received BRV 50 mg/day during 2 weeks of Transition Period and BRV 100 mg/day in LTFU study or MAP. Participants who did not enter the LTFU study or MAP had 4 weeks Down-Titration Period followed by a Study Drug-Free Period (no drug for 2 weeks). During Down-Titration Period, participants received BRV 25 mg/day for 1 week followed by Placebo for 3 weeks.
- BRV 200 mg/Day: Participants received BRV 200 mg/day as film-coated tablets, administered orally, bid, during 12 weeks of Treatment Period. At the end of the Treatment Period, participants who entered LTFU study or MAP received BRV 150 mg/day during 2 weeks of Transition Period and BRV 100 mg/day in LTFU study or MAP. Participants who did not enter the LTFU study or MAP had 4 weeks Down-Titration Period followed by a Study Drug-Free Period (no drug for 2 weeks). During Down-Titration Period, participants received BRV 150 mg/day for 1 week followed by BRV 100 mg/day for 1 week, followed by BRV 50 mg/day for 1 week, followed by BRV 25 mg/day for 1 week.
- Placebo to OLTP BRV: Participants who received Placebo during Treatment Period and were eligible to enter MAP received BRV 100 mg/day due to delayed importation of medication during OLTP. BRV dose might be adjusted for an individual participant (between 50 mg/day to 200 mg/day) during the OLTP. The period was defined from immediately after the last visit of the Transition Period (Week 14) and until a visit when the participant could convert to MAP.
- BRV 50 mg/Day to OLTP BRV: Participants who received BRV 50 mg/day during Treatment Period and were eligible to enter MAP received BRV 100 mg/day due to delayed importation of medication during Open-Label Temporary Period (OLTP). BRV dose might be adjusted for an individual participant (between 50 mg/day to 200 mg/day) during the OLTP. The period was defined from immediately after the last visit of the Transition Period (Week 14) and until a visit when the participant could convert to MAP.
- BRV 200 mg/Day to OLTP BRV: Participants who received BRV 200 mg/day during Treatment Period and were eligible to enter MAP received BRV 100 mg/day due to delayed importation of medication during Open-Label Temporary Period (OLTP). BRV dose might be adjusted for an individual participant (between 50 mg/day to 200 mg/day) during the OLTP. The period was defined from immediately after the last visit of the Transition Period (Week 14) and until a visit when the participant could convert to MAP.
Period: Double-Blind Period
Arm/Group | Placebo | BRV 50 mg/Day | BRV 200 mg/Day | Placebo to OLTP BRV | BRV 50 mg/Day to OLTP BRV | BRV 200 mg/Day to OLTP BRV
Started | 149 | 152 | 148 | 0 | 0 | 0
Started Treatment Period (12 Weeks) | 149 | 152 | 148 | 0 | 0 | 0
Started Down-Titration Period (4 Weeks) | 7 | 9 | 7 | 0 | 0 | 0
Started Study Drug-Free Period (2 Weeks) | 7 | 9 | 7 | 0 | 0 | 0
Started Transition Period (2 Weeks) | 133 | 139 | 137 | 0 | 0 | 0
Completed | 138 | 147 | 140 | 0 | 0 | 0
Not Completed | 11 | 5 | 8 | 0 | 0 | 0
Not completed — Adverse Event | 5 | 4 | 5 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Consent withdrawn by subject due to concern on AE | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Subjects were able to never take a study drug | 0 | 1 | 0 | 0 | 0 | 0
Period: Open-Label Temporary Period (OLTP)
Arm/Group | Placebo | BRV 50 mg/Day | BRV 200 mg/Day | Placebo to OLTP BRV | BRV 50 mg/Day to OLTP BRV | BRV 200 mg/Day to OLTP BRV
Started | 0 | 0 | 0 | 64 | 68 | 74
Completed | 0 | 0 | 0 | 60 | 67 | 68
Not Completed | 0 | 0 | 0 | 4 | 1 | 6
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 1 | 1
Not completed — Withdrawal by parent/guardian | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Patient not keen to continue open label | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Patient non compliant to open label study drug | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Subject enrolled to compassionate use program | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Randomized Set (RS) which consisted of all study participants who were randomized to investigational medicinal product (IMP).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BRV 50 mg/Day | BRV 200 mg/Day | Total
Number analyzed (Participants) | 149 | 152 | 148 | 449
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 14 | 8 | 31
  Between 18 and 65 years | 137 | 135 | 138 | 410
  >=65 years | 3 | 3 | 2 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (13.2) | 33.7 (12.6) | 35.2 (13.2) | 34.5 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 77 | 83 | 242
  Male | 67 | 75 | 65 | 207
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 149 | 152 | 148 | 449
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 3
  Not Hispanic or Latino | 148 | 151 | 147 | 446

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An AE is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. Treatment-Emergent AEs were defined as AEs which had onset on or after the first dose of IMP. As per planned analysis, safety data for all study periods was combined excluding Open-Label Temporary period.
Time Frame: From start of the Treatment Period (Week 0) until Safety Visit (up to Week 18); only for OLTP- From last visit of Transition Period to beginning of MAP (up to 4 Years 10 Months)
Population: The Safety Set (SS) included all randomized study participants who received at least 1 dose of IMP.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | BRV 50 mg/Day | BRV 200 mg/Day | Placebo to OLTP BRV | BRV 50 mg/Day to OLTP BRV | BRV 200 mg/Day to OLTP BRV
Number analyzed (Participants) | 149 | 151 | 148 | 64 | 68 | 74
percentage of participants | 58.4 | 57.0 | 60.1 | 26.6 | 19.1 | 23.0

2. Primary Outcome: Percentage of Participants With Treatment-Emergent AEs (TEAEs) Leading to Study Withdrawal
Description: as for outcome 1
Time Frame: as for outcome 1
Population: The SS included all randomized study participants who received at least 1 dose of IMP.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | BRV 50 mg/Day | BRV 200 mg/Day | Placebo to OLTP BRV | BRV 50 mg/Day to OLTP BRV | BRV 200 mg/Day to OLTP BRV
Number analyzed (Participants) | 149 | 151 | 148 | 64 | 68 | 74
percentage of participants | 4.7 | 2.6 | 3.4 | 0 | 0 | 0

3. Primary Outcome: Percentage of Participants With Treatment-Emergent Serious Adverse Events (SAEs)
Description: Serious Adverse event (SAE) was defined as any events which: • results in death, • is life-threatening threatening (note that this did not include a reaction that might have caused death had it occurred in a more severe form.), •results in significant or persistent disability/incapacity, • results in a congenital anomaly/birth defect (including that occurring in a fetus), • results in Important medical event that, based upon appropriate medical judgment, may jeopardize the participant and might require medical or surgical intervention to prevent 1 of the other outcomes listed here, and • results in initial inpatient hospitalization or prolongation of hospitalization. As per planned analysis, safety data for all study periods was combined excluding Open-Label Temporary period.
Time Frame: as for outcome 1
Population: The SS included all randomized study participants who received at least 1 dose of IMP.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | BRV 50 mg/Day | BRV 200 mg/Day | Placebo to OLTP BRV | BRV 50 mg/Day to OLTP BRV | BRV 200 mg/Day to OLTP BRV
Number analyzed (Participants) | 149 | 151 | 148 | 64 | 68 | 74
percentage of participants | 0.7 | 1.3 | 2.7 | 4.7 | 0 | 2.7

4. Primary Outcome: Partial Seizure Frequency Per 28 Days During the 12-week Treatment Period
Description: According to International League Against Epilepsy (ILAE) classification (1981), seizures were classified as type IA (IA1, IA2, IA3, and IA4), IB, IC, II (IIA, IIB, IIC, IID, IIE, and IIF) or III. 28 day adjusted seizure frequency for partial seizures (seizure types IA+IB+IC) was calculated for treatment period by dividing the number of partial seizures by the number of days for which the DRC was completed for treatment period and multiplying the resulting value by 28.
Time Frame: From Baseline to 12-week Treatment Period
Population: The Full Analysis Set (FAS) consisted of all randomized study participants who received at least 1 dose of IMP and had at least 1 post Baseline seizure daily record card (DRC) data during the Treatment Period.
Measure: Median (Full Range); unit: seizures per 28 days
Arm/Group | Placebo | BRV 50 mg/Day | BRV 200 mg/Day
Number analyzed (Participants) | 147 | 151 | 148
seizures per 28 days | 7.17 [1.0 to 317.0] | 5.93 [0.0 to 123.7] | 4.19 [0.0 to 269.4]
Statistical Analysis 1: Comparison: Placebo vs BRV 50 mg/Day; Test type: Superiority; p = 0.0005, ANCOVA — Statistical testing with control of Type I error rate were based on a Hochberg multiple comparison procedure; Percent reduction over Placebo = 24.5, 95% CI 2-sided [11.7 to 35.5] — Based on ANCOVA with log-transformed [log(x+1)] Treatment Period 28-day adjusted partial seizure frequency
Statistical Analysis 2: Comparison: Placebo vs BRV 200 mg/Day; Test type: Superiority; p < 0.0001, ANCOVA — Statistical testing with control of Type I error rate were based on a Hochberg multiple comparison procedure; Percent reduction over Placebo = 33.4, 95% CI 2-sided [21.9 to 43.1] — Based on ANCOVA with log-transformed [log(x+1)] Treatment Period 28-day adjusted partial seizure frequency

5. Secondary Outcome: 50% Responder Rate Based on Percent Change in Partial Seizure Frequency Per 28 Days From Baseline to the 12-week Treatment Period
Description: Responders were those participants with at least 50% reduction from Baseline to the 12-week Treatment Period in partial seizure frequency per 28 days. 50% Responder rate was calculated for treatment period by dividing the number of 50% responders by the number of participants in the analysis set and multiplying the resulting value by 100.
Time Frame: From Baseline to 12-week Treatment Period
Population: The FAS consisted of all randomized study participants who received at least 1 dose of IMP and had at least 1 post Baseline seizure DRC data during the Treatment Period.
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Placebo | BRV 50 mg/Day | BRV 200 mg/Day
Number analyzed (Participants) | 147 | 151 | 148
percentage of responders | 19.0 [13.0 to 26.3] | 41.1 [33.1 to 49.3] | 49.3 [41.0 to 57.7]

6. Secondary Outcome: Percent Change in Partial Seizure Frequency Per 28 Days From Baseline to the 12-week Treatment Period
Description: Percent change from Baseline to the Treatment Period in partial seizure frequency was calculated by subtracting 28-day adjusted Treatment Period partial seizure frequency from 28-day adjusted Baseline Period partial seizure frequency, and multiplying the resulting quantity by 100 and dividing by the Baseline Period 28-day adjusted partial seizure frequency. A negative value in percent change from Baseline indicates a decrease in partial seizure frequency from Baseline to the Treatment Period.
Time Frame: From Baseline to 12-week Treatment Period
Population: as for outcome 5
Measure: Median (Full Range); unit: percent change
Arm/Group | Placebo | BRV 50 mg/Day | BRV 200 mg/Day
Number analyzed (Participants) | 147 | 151 | 148
percent change | 21.3 [-123 to 87] | 38.9 [-233 to 100] | 46.7 [-1097 to 100]

7. Secondary Outcome: Percentage of Participants With Categorized Percent Change in Partial Seizure Frequency Per 28 Days From Baseline to the 12-week Treatment Period
Description: The percentage of participants within each of the following categories of percent change in partial seizure frequency from Baseline to the Treatment Period were summarized for each treatment group: 100%, 75% to less than 100%, 50% to less than 75%, 25% to less than 50%, -25% to less than 25%, and less than -25%. Percent change from Baseline to the Treatment Period in partial seizure frequency was calculated by subtracting 28-day adjusted Treatment Period partial seizure frequency from 28-day adjusted Baseline Period partial seizure frequency and multiplying the resulting quantity by 100 and dividing by the Baseline Period 28-day adjusted partial seizure frequency.
Time Frame: From Baseline to 12-week Treatment Period
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | BRV 50 mg/Day | BRV 200 mg/Day
Number analyzed (Participants) | 147 | 151 | 148
percentage of participants
  100% | 0 | 5.3 | 7.4
  75% to less than 100% | 3.4 | 14.6 | 17.6
  50% to less than 75% | 15.6 | 21.2 | 24.3
  25% to less than 50% | 27.2 | 16.6 | 20.9
  -25% to less than 25% | 42.9 | 31.1 | 18.2
  less than-25% | 10.9 | 11.3 | 11.5

8. Secondary Outcome: All Seizure Frequency (Partial, Generalized, and Unclassified Epileptic Seizures) Per 28 Days During the 12-week Treatment Period
Description: There were three types of epileptic seizures: Partial epileptic seizures (Type I), Generalized epileptic seizures (Type II) and unclassified epileptic seizures (Type III). 28 day adjusted seizure frequency for all seizure types was calculated for treatment period by dividing the number of targeted seizures by the number of days for which the DRC was completed for treatment period and multiplying the resulting value by 28.
Time Frame: During the 12-week Treatment Period
Population: as for outcome 5
Measure: Median (Full Range); unit: seizures per 28 days
Arm/Group | Placebo | BRV 50 mg/Day | BRV 200 mg/Day
Number analyzed (Participants) | 147 | 151 | 148
seizures per 28 days | 7.17 [1.0 to 317.0] | 5.93 [0.0 to 123.7] | 4.19 [0.0 to 269.4]

9. Secondary Outcome: Percentage of Participants Who Are Seizure Free (Partial, All Epileptic Seizures) During the 12-week Treatment Period
Description: Participants were defined as seizure free, if they did not have missing diary days and no reported seizures during the Treatment Period.
Time Frame: During the 12-week Treatment Period
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | BRV 50 mg/Day | BRV 200 mg/Day
Number analyzed (Participants) | 147 | 151 | 148
percentage of participants
  All epileptic seizures | 0 | 4.6 | 6.8
  Partial onset seizures | 0 | 4.6 | 6.8

10. Secondary Outcome: Time to 1st Partial Seizure During the 12-week Treatment Period
Description: The evaluation of time to 1st partial seizure was based on the relative day of occurrence of the 1st partial seizure during the Treatment Period.
Time Frame: During the 12-week Treatment Period
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | BRV 50 mg/Day | BRV 200 mg/Day
Number analyzed (Participants) | 147 | 151 | 148
days | 3 [2 to 3] | 5 [3 to 6] | 6 [5 to 8]

11. Secondary Outcome: Time to 5th Partial Seizure During the 12-week Treatment Period
Description: The evaluation of time to 5th partial seizure was based on the relative day of occurrence of the 5th partial seizure during the Treatment Period.
Time Frame: During the 12-week Treatment Period
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | BRV 50 mg/Day | BRV 200 mg/Day
Number analyzed (Participants) | 147 | 151 | 148
days | 17 [15 to 21] | 28 [23 to 36] | 32 [29 to 38]

12. Secondary Outcome: Time to 10th Partial Seizure During the 12-week Treatment Period
Description: The evaluation of time to 10th partial seizure was based on the relative day of occurrence of the 10th partial seizure during the Treatment Period.
Time Frame: During the 12-week Treatment Period
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | BRV 50 mg/Day | BRV 200 mg/Day
Number analyzed (Participants) | 147 | 151 | 148
days | 43 [32 to 52] | 59 [48 to 76] | 69 [59 to NA] — Upper limit of 95% Confidence interval (CI) was not calculated due to less number of participants with events.

13. Secondary Outcome: Brivaracetam Plasma Concentration
Description: Blood samples were collected at indicated time points for the 50mg/day and 200mg/day groups to determine the brivaracetam plasma concentration. Participants of arm 'BRV 200 mg/day' received BRV 200 mg/day until Week 12 only and 150 mg/day during the Transition Period at Week 14. Therefore, the data is reported according to the dosage information at specified time point. As per planned analysis, one blood sample was collected for BRV plasma levels during each dosing interval between 0 to 4 hours, 4 to 8 hours, and 8 to 12 hours postdose.
Time Frame: Plasma samples were collected at >0-4hours, >4-8hours, >8hours in weeks 2, 4, 8, 12, and 14
Population: The Pharmacokinetic Per-Protocol Set (PK-PPS) consisted of all study participants who took at least 1 dose of BRV and for whom at least 1 valid BRV plasma concentration time and dosing information were available. Here, 'n' (Number analyzed) signifies participants who were evaluable at specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/ millilitre (ug/mL)
Groups:
- BRV 150 mg/Day: At the end of the Treatment Period, participants of arm BRV 200 mg/day who entered LTFU study or MAP received BRV 150 mg/day during 2 weeks of Transition Period. The number of participants for BRV 150 mg/day group are those who had BRV 200 mg/day and valid PK data in Transition Period.
Arm/Group | BRV 50 mg/Day | BRV 200 mg/Day | BRV 150 mg/Day
Number analyzed (Participants) | 150 | 146 | 128
microgram/ millilitre (ug/mL)
  Week 2: > 0 - 4 hours: number analyzed (Participants) | 120 | 99 | 0
  Week 2: > 0 - 4 hours | 0.68556 (95.6) | 3.4340 (42.5) |
  Week 2: > 4 - 8 hours: number analyzed (Participants) | 18 | 27 | 0
  Week 2: > 4 - 8 hours | 0.66523 (38.6) | 2.0615 (334.4) |
  Week 2: > 8 hours: number analyzed (Participants) | 8 | 15 | 0
  Week 2: > 8 hours | 0.18427 (979.4) | 1.2144 (100.1) |
  Week 4: > 0 - 4 hours: number analyzed (Participants) | 118 | 101 | 0
  Week 4: > 0 - 4 hours | 0.75902 (88.8) | 3.0038 (120.2) |
  Week 4: > 4 - 8 hours: number analyzed (Participants) | 18 | 31 | 0
  Week 4: > 4 - 8 hours | 0.64781 (39.2) | 2.8516 (43.2) |
  Week 4: > 8 hours: number analyzed (Participants) | 7 | 7 | 0
  Week 4: > 8 hours | 0.39652 (54.7) | 1.1054 (74.4) |
  Week 8: > 0 - 4 hours: number analyzed (Participants) | 115 | 146 | 0
  Week 8: > 0 - 4 hours | 0.76942 (87.3) | 2.9983 (127.7) |
  Week 8: > 4 - 8 hours: number analyzed (Participants) | 19 | 24 | 0
  Week 8: > 4 - 8 hours | 0.76172 (34.0) | 2.7030 (54.9) |
  Week 8: > 8 hours: number analyzed (Participants) | 7 | 9 | 0
  Week 8: > 8 hours | 0.27840 (10.9) | 1.5590 (67.7) |
  Week 12: > 0 - 4 hours: number analyzed (Participants) | 98 | 97 | 0
  Week 12: > 0 - 4 hours | 0.77400 (89.5) | 3.2508 (121.1) |
  Week 12: > 4 - 8 hours: number analyzed (Participants) | 28 | 29 | 0
  Week 12: > 4 - 8 hours | 0.65274 (39.4) | 1.6017 (838.9) |
  Week 12: > 8 hours: number analyzed (Participants) | 10 | 9 | 0
  Week 12: > 8 hours | 0.18229 (579.5) | 1.5001 (45.4) |
  Week 14 (Transition): > 0 - 4 hours: number analyzed (Participants) | 106 | 0 | 95
  Week 14 (Transition): > 0 - 4 hours | 0.75949 (85.3) |  | 2.4989 (54.8)
  Week 14 (Transition): > 4 - 8 hours: number analyzed (Participants) | 15 | 0 | 28
  Week 14 (Transition): > 4 - 8 hours | 0.75692 (34.6) |  | 1.4383 (309.5)
  Week 14 (Transition): > 8 hours: number analyzed (Participants) | 7 | 0 | 5
  Week 14 (Transition): > 8 hours | 0.41286 (66.4) |  | 0.82681 (30.6)

ADVERSE EVENTS:
Time Frame: From start of the Treatment Period (Week 0) until Safety Visit (up to Week 18); only for OLTP- From last visit of Transition Period to beginning of MAP (Up to 4 Years 10 Months)
Description: TEAEs were defined as AEs which had onset on or after the first dose of investigational medicinal product (IMP). The Safety Set (SS) included all randomized participants who took at least 1 dose of study medication. As per planned analysis, safety data for all study periods was combined excluding Open-Label Temporary period.
Arm/Group | Placebo | BRV 50 mg/Day | BRV 200 mg/Day | Placebo to OLTP BRV | BRV 50 mg/Day to OLTP BRV | BRV 200 mg/Day to OLTP BRV
All-Cause Mortality (participants affected / at risk) | 0/149 | 1/151 | 0/148 | 0/64 | 0/68 | 0/74
Serious Adverse Events (participants affected / at risk) | 1/149 | 2/151 | 4/148 | 3/64 | 0/68 | 2/74
Other Adverse Events (participants affected / at risk) | 39/149 | 42/151 | 54/148 | 3/64 | 4/68 | 4/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=149) | BRV 50 mg/Day (N=151) | BRV 200 mg/Day (N=148) | Placebo to OLTP BRV (N=64) | BRV 50 mg/Day to OLTP BRV (N=68) | BRV 200 mg/Day to OLTP BRV (N=74)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drowning (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Corona virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postictal psychosis (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Miscarriage of partner (Social circumstances) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Near drowning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cervicogenic headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=149) | BRV 50 mg/Day (N=151) | BRV 200 mg/Day (N=148) | Placebo to OLTP BRV (N=64) | BRV 50 mg/Day to OLTP BRV (N=68) | BRV 200 mg/Day to OLTP BRV (N=74)
Upper respiratory tract infection (Infections and infestations) | 7 (8) | 10 (14) | 8 (9) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 10 (11) | 7 (10) | 10 (10) | 3 (3) | 4 (5) | 4 (4)
Somnolence (Nervous system disorders) | 12 (14) | 15 (15) | 28 (29) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 6 (6) | 17 (19) | 21 (24) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 11 (15) | 11 (16) | 7 (8) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-01-10): https://cdn.clinicaltrials.gov/large-docs/65/NCT03083665/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-17): https://cdn.clinicaltrials.gov/large-docs/65/NCT03083665/SAP_001.pdf